CLINICAL TRIAL: NCT01325207
Title: Phase I/II Dose Escalation Trial to Assess Safety of Intrathecal Trastuzumab for the Treatment of Leptomeningeal Metastases in HER2 Positive Breast Cancer
Brief Title: Intrathecal Trastuzumab for Leptomeningeal Metastases in HER2+ Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 10C03; STU00040150 (Other: Northwestern University IRB)
Record Dates: First submitted 2011-03-07; First posted 2011-03-29 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intravenous trastuzumab infusions (Experimental): A Phase I single dose study (H0407g) of intravenous trastuzumab infusions ranging from 10-500 mg resulted in dose-dependent pharmacokinetics (PK) with serum clearance of trastuzumab decreasing with an increasing dose at doses <250 mg. PK modeling of trastuzumab concentration-time data from 7 patients that were administered doses of 250 mg and 500 mg had in a mean halflife of 5.8 days (range 1-32 days).
  Interventions: Radiation: Trastuzumab

INTERVENTIONS:
Radiation: Trastuzumab — Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks
  Other Names: (also known as Herceptin, which; is a medicine that is used to slow or stop the growth of a cancerous tumor)

SUMMARY:
The drug being studied is Trastuzumab, a medicine that is used to slow or stop the growth of cancerous tumors that are HER-2 positive. Patients are being asked to participate in this study because they have been diagnosed with having tumor cells in their spinal fluid. This study will investigate the safety and effects of this drug when given directly into the spinal fluid.

Phase I/II Dose Escalation Trial to Assess Safety of Intrathecal Trastuzumab for the Treatment of Leptomeningeal Metastases in HER2 Positive Breast Cancer The purpose of this research study is to determine a safe dose of the drug Trastuzumab and then determine how effective this treatment is.

DETAILED DESCRIPTION:
Phase I: Patients will be treated in cohorts of 3-6 based on standard phase I dose escalation parameters requiring 0/3 or 1/6 patients per cohort to have a DLT before dose escalation. Dosing is as follows: Cohort 1-10 mg IT, cohort 2-20 mg IT, cohort 3-30 mg IT and cohort 4-40 mg IT. Patients will be treated twice a week for 4 weeks, then once a week for 4 weeks, and then every 2 weeks. Toxicity for DLT will be assessed during first 4 weeks of treatment. Phase II: Patients will be treated with the MTD or maximal defined dose. Patients will be treated twice a week for 4 weeks, then once a week for 4 weeks, and then every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

ELIGIBILITY CRITERIA

* HER2 positive (IHC 3+ and/or FISH positive) breast cancer patients with leptomeningeal metastases by MRI or CSF (if MRI is negative).

  o Review will be performed for cases not reviewed at Northwestern for confirmation, but will not preclude patients from entering the trial (pathology report is sufficient for registration).
* Patients can have concomitant brain metastases as long as they do not require active treatment or have been treated.
* Patients with leptomeningeal disease from ependymomas, gliomas, and medulloblastoma will be eligible for phase I
* Life expectancy > 8 weeks
* Normal renal (creatinine < 1.5 ULN), liver (bilirubin < 1.5 x ULN, transaminases < 3.0 x ULN, except in known hepatic metastasis, wherein may be < 5 x ULN) and blood counts (WBC > 3.0, Neutrophils > 1500, platelets >100 000, Hemoglobin > 10).
* LVEF > 50%
* KPS > 50
* Age > 18 years
* Cannot be on systemic agents (chemotherapy) that have CNS penetration unless they develop leptomeningeal metastases while on these agent(s) and have controlled systemic disease. May continue on IV trastuzumab, lapatinib or hormonal agents if controlling systemic disease and developed LM while on therapy. Patients requiring systemic chemotherapy are eligible but will not be able to start treatment until after the first assessment by imaging and cytology.
* Patients may need a CSF flow study at the discretion of the treating principal investigator. If a spinal block is seen by CSF flow study or MRI, it will need local RT prior to treatment. Concurrent radiation is not allowed.
* Patients should be > 2 weeks from RT treatment and all effects of treatment should have resolved
* No limit on prior systemic or IT therapies.
* CSF sampling to document LM if not documented on MRI.
* Must be willing to have an Ommaya reservoir placed.
* NO history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless in complete remission and off all therapy for the disease for a minimum of 3 years.
* Significant medical or psychiatric illness that would interfere with compliance and ability to tolerate treatment as outlined in the protocol.
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study.
* Women may not be pregnant or breast-feeding.
* Ability to sign an informed consent; can be signed by family member or health care proxy. Informed consent must be done prior to registration on study.
* All patients must have given signed, informed consent prior to registration on study.
* No known hypersensitivity to trial medications Note: The eligibility criteria listed above are interpreted literally and cannot be waived.

Exclusion Criteria:

- Any deviations from the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-08-01; Primary Completion 2016-06-20 (Actual); Study Completion 2019-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Raizer, MD, Principal Investigator — Northwestern University
Locations (8):
- United States (8):
  - University of California San Francisco (UCSF), San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - Texas Oncology-Austin, Austin, Texas

REFERENCES:
- [Derived] Malani R, Fleisher M, Kumthekar P, Lin X, Omuro A, Groves MD, Lin NU, Melisko M, Lassman AB, Jeyapalan S, Seidman A, Skakodub A, Boire A, DeAngelis LM, Rosenblum M, Raizer J, Pentsova E. Cerebrospinal fluid circulating tumor cells as a quantifiable measurement of leptomeningeal metastases in patients with HER2 positive cancer. J Neurooncol. 2020 Jul;148(3):599-606. doi: 10.1007/s11060-020-03555-z. Epub 2020 Jun 6. PMID 32506369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on April 26, 2011 with first patient being treated August 1, 2011, with an accrual goal of up to 48 patients for phase I/II combined. Amendment 5 added 5th cohort to allow higher dose. The study was suspended April 12, 2014 and reopened on August 28, 2014 for phase II. The study closed to accrual June 2, 2016.
Groups:
- Cohort 1 - Trastuzumab 10mg IT 2/Week: Intrathecal Trastuzumab 10 mg IT will be administered in Cohort 1 of dose escalation.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks until disease progression or unacceptable toxicity.
  1 cycle = 28 days.
- Cohort 2 - Trastuzumab 20mg IT 2/Week: Intrathecal Trastuzumab 20 mg IT will be administered in Cohort 2 of dose escalation.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks until disease progression or unacceptable toxicity.
  1 cycle = 28 days.
- Cohort 3- Trastuzumab 40mg IT 2/Week: Intrathecal Trastuzumab 40 mg IT will be administered in Cohort 3 of dose escalation.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks until disease progression or unacceptable toxicity.
  1 cycle = 28 days.
- Cohort 4 - Trastuzumab 60mg IT 2/Week: Intrathecal Trastuzumab 60 mg IT will be administered in Cohort 4 of dose escalation.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks until disease progression or unacceptable toxicity.
  1 cycle = 28 days.
- Cohort 5 - 80mg IT 2/Week: Intrathecal Trastuzumab 80 mg IT will be administered in Cohort 5 of dose escalation.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks until disease progression or unacceptable toxicity.
  1 cycle = 28 days.
- Phase II - Transtuzumab 80mg IT 2/Week: Intrathecal Trastuzumab 10 mg IT will be administered in phase II portion of the study.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks until disease progression or unacceptable toxicity.
  1 cycle = 28 days.
Period: Completed 4 Weeks/1 Cycle of Treatment
Arm/Group | Cohort 1 - Trastuzumab 10mg IT 2/Week | Cohort 2 - Trastuzumab 20mg IT 2/Week | Cohort 3- Trastuzumab 40mg IT 2/Week | Cohort 4 - Trastuzumab 60mg IT 2/Week | Cohort 5 - 80mg IT 2/Week | Phase II - Transtuzumab 80mg IT 2/Week
Started | 3 | 3 | 1 | 1 | 7 | 19
Completed | 3 | 3 | 1 | 1 | 5 | 19
Not Completed | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0
Period: Completed 8 Weeks/2 Cycles of Treatment
Arm/Group | Cohort 1 - Trastuzumab 10mg IT 2/Week | Cohort 2 - Trastuzumab 20mg IT 2/Week | Cohort 3- Trastuzumab 40mg IT 2/Week | Cohort 4 - Trastuzumab 60mg IT 2/Week | Cohort 5 - 80mg IT 2/Week | Phase II - Transtuzumab 80mg IT 2/Week
Started | 3 | 3 | 1 | 1 | 5 | 19
Completed | 2 | 2 | 1 | 1 | 3 | 14
Not Completed | 1 | 1 | 0 | 0 | 2 | 5
Not completed — Progressive Disease | 1 | 1 | 0 | 0 | 2 | 5
Period: Started 9th Week/Cycle 3 of Treatment
Arm/Group | Cohort 1 - Trastuzumab 10mg IT 2/Week | Cohort 2 - Trastuzumab 20mg IT 2/Week | Cohort 3- Trastuzumab 40mg IT 2/Week | Cohort 4 - Trastuzumab 60mg IT 2/Week | Cohort 5 - 80mg IT 2/Week | Phase II - Transtuzumab 80mg IT 2/Week
Started | 2 | 2 | 1 | 1 | 3 | 14
Completed | 1 | 0 | 0 | 0 | 3 | 9
Not Completed | 1 | 2 | 1 | 1 | 0 | 5
Not completed — Progressive disease | 1 | 1 | 1 | 1 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Follow-up Every 3 Months Until Death
Arm/Group | Cohort 1 - Trastuzumab 10mg IT 2/Week | Cohort 2 - Trastuzumab 20mg IT 2/Week | Cohort 3- Trastuzumab 40mg IT 2/Week | Cohort 4 - Trastuzumab 60mg IT 2/Week | Cohort 5 - 80mg IT 2/Week | Phase II - Transtuzumab 80mg IT 2/Week
Started (All patients treated on study went into the follow up period.) | 3 | 3 | 1 | 1 | 7 | 19
Completed | 3 | 3 | 1 | 1 | 6 | 18
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Follow-up Considered Complete | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Trastuzumab 10mg IT 2/Week | Cohort 2 - Trastuzumab 20mg IT 2/Week | Cohort 3- Trastuzumab 40mg IT 2/Week | Cohort 4 - Trastuzumab 60mg IT 2/Week | Cohort 5 - 80mg IT 2/Week | Phase II - Transtuzumab 80mg IT 2/Week | Total
Number analyzed (Participants) | 3 | 3 | 1 | 1 | 7 | 19 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 1 | 1 | 6 | 17 | 31
  >=65 years | 0 | 0 | 0 | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 1 | 7 | 18 | 32
  Male | 1 | 0 | 0 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 2 | 3 | 1 | 1 | 7 | 18 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 3 | 3
  White | 3 | 3 | 1 | 1 | 7 | 14 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 1 | 1 | 7 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLT) of IT Trastuzumab in Sequential Cohorts of Escalating Doses for Patients With Leptomeningeal Metastases in HER2+ Breast Cancer.
Description: Patients will be treated using a standard 3+3 dose-escalation design for cohorts 1 and 2. This will be followed by an accelerated phase I for cohorts 3 and 4, and then a standard 3 + 3 for the 5th cohort. In the accelerated phase (cohorts 3 and 4), 1 patient will be enrolled per cohort; if a toxicity is seen in that patient then the cohort would be expanded to 6 patients to allow for 1/6 patients per cohort to have a dose limiting toxicity (DLT) before dose escalation. Cohort 5 will enroll a total of 6 patients regardless of the toxicity experienced in patient one. However, if 2 or more DLTs are observed in cohort 5, cohort 4 will be reopened to enroll of a total of 6 patients. Whatever dose is ultimately declared the MTD should have 6 patients total. If 1/6 DLTs are seen in cohort 5 that will be considered the MTD.
  Dosing is as follows:
  Cohort 1-10 mg IT Cohort 2-20 mg IT Cohort 3-40 mg IT Cohort 4-60 mg IT Cohort 5-80 mg IT
Time Frame: From treatment initiation through the first 4 weeks of treatment.
Measure: Number; unit: DLTs
Arm/Group | Cohort 1 - Trastuzumab 10mg IT 2/Week | Cohort 2 - Trastuzumab 20mg IT 2/Week | Cohort 3- Trastuzumab 40mg IT 2/Week | Cohort 4 - Trastuzumab 60mg IT 2/Week | Cohort 5 - 80mg IT 2/Week
Number analyzed (Participants) | 3 | 3 | 1 | 1 | 7
DLTs | 0 | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Cohort 1 - Trastuzumab 10mg IT 2/Week vs Cohort 2 - Trastuzumab 20mg IT 2/Week vs Cohort 3- Trastuzumab 40mg IT 2/Week vs Cohort 4 - Trastuzumab 60mg IT 2/Week vs Cohort 5 - 80mg IT 2/Week; Test type: Other; The Maximum Tolerated Dose (MTD) was determined to be 80mg IT every two weeks. This is based on no DLTs being seeing in Cohorts 1-4 with lower doses and 1 DLT out of 7 patients observed at 80mg IT in Cohort 5

2. Primary Outcome: Best Response to IT Trastuzumab: Radiological, Cytological and Clinical in Treatment With Intrathecal Trastuzumab for Patients With Leptomeningeal Metastases in HER2+ Breast Cancer.
Description: Best response will be assessed using a combination CSF cytology assessment, radiographic assessment and clinical function assessments. Best response will be defined as the best response seen during treatment as compared to baseline that is confirmed on subsequent response assessment.
Time Frame: Baseline then at 4 weeks, 8 weeks and then every 8 weeks +/- 3 days, until disease progression or toxicity,range of cycles completed 1-22 cycles where 1 cycle = 28 days.
Population: All patients were assessed for response. Patients unable to be assessed were determined to have progressive disease and counted. Cohort results for this outcome measure were analysed combined and at the MTD of 80mg IT (Cohort 5 + phase II). The objective was to determine preliminary response data for this treatment combination.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment With Trastuzumab: Intrathecal Trastuzumab will be administered in a dose escalation design from 10mg up to 80 mg IT.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks.
  1 cycle = 28 days
- Cohort 5 + Phase II - Intrathecal Trastuzumab- 80 mg: Intrathecal Trastuzumab will be administered at the MTD determined dose of 80 mg IT.
  Trastuzumab: Trastuzumab will be administered twice per week for 4 weeks, then once per week for 4 weeks, and then every 2 weeks.
  1 cycle = 28 days
Arm/Group | Treatment With Trastuzumab | Cohort 5 + Phase II - Intrathecal Trastuzumab- 80 mg
Number analyzed (Participants) | 34 | 26
Participants
  Complete Response | 0 | 0
  Partial Response | 6 | 5
  Stable Disease | 18 | 13
  Progressive Disease | 10 | 8

3. Other Pre Specified Outcome: Define the CSF PK of IT Trastuzumab.
Description: Patients may need a CSF flow study at the discretion of the treating principal investigator. If a spinal block is seen by CSF flow study or MRI, it will need local RT prior to treatment. Concurrent radiation is not allowed.
Time Frame: CSF analysis for cytology will be done every 2 weeks when CSF is obtained for PK and then every 4 weeks
Reporting Status: Not Posted

4. Post Hoc Outcome: Progression Free Survival (PRS) at 6 Months and at 12 Months in Treatment With Intrathecal Trastuzumab for Patients With Leptomeningeal Metastases in HER2+ Breast Cancer.
Description: Progression Free Survival (PFS) will be measured from the time of treatment initiation until the first documentation of progression. To estimate the probability of PFS at 6 months and 12 months, Kaplan-Meier curves will be calculated and PFS at 6 months and 12 months will be determined from the progression-free survival curve. Progression will be defined as worsening clinical signs or development of new clinical symptoms that the Investigator feels can be attributed to Leptomeningeal disease.
Time Frame: At 6 and 12 months from start of treatment
Population: Cohort results for this outcome measure were analyzed both combined and for patients treated at the MTD dose of 80mg IT as the objective was to determine preliminary data on PFS of patients with this drug combination.
Measure: Number; unit: Probability of Survival
Arm/Group | Treatment With Trastuzumab | Cohort 5 + Phase II - Intrathecal Trastuzumab- 80 mg
Number analyzed (Participants) | 34 | 26
Probability of Survival
  PFS at 6 months | 0.235 | 0.269
  PFS at 12 months | 0.118 | 0.115

5. Post Hoc Outcome: Overall Survival (OS) at 6 and 12 Months in Treatment With Intrathecal Trastuzumab for Patients With Leptomeningeal Metastases in HER2+ Breast Cancer.
Description: Overall Survival (OS) will be measured from the time of treatment initiation until death from any cause. To estimate OS probability at 6 and 12 months, Kaplan-Meier curves will be calculated and OS at 612 months will be determined from the overall survival curve.
Time Frame: At 6 and 12 months from start of treatment
Population: Cohort results for this outcome measure were analyzed both combined and for patients treated at the MTD dose of 80mg IT as the objective was to determine preliminary data on OS of patients with this drug combination.
Measure: Number; unit: Probability of Survival
Arm/Group | Treatment With Trastuzumab | Cohort 5 + Phase II - Intrathecal Trastuzumab- 80 mg
Number analyzed (Participants) | 34 | 26
Probability of Survival
  OS at 6 months | 0.562 | 0.542
  OS at 12 months | 0.406 | 0.458

6. Post Hoc Outcome: Median Progression Free Survival (PFS) in Treatment With Intrathecal Trastuzumab for Patients With Leptomeningeal Metastases in HER2+ Breast Cancer.
Description: Progression Free Survival (PFS) will be measured from the time of treatment initiation until the first documentation of progression. To estimate PFS, Kaplan-Meier curves will be calculated and the median PFS will be determined from the progression-free survival curve. Progression will be defined as worsening clinical signs or development of new clinical symptoms that the Investigator feels can be attributed to Leptomeningeal disease.
Time Frame: From start of treatment, and during treatment until progressive disease for up to 30 months.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment With Trastuzumab | Cohort 5 + Phase II - Intrathecal Trastuzumab- 80 mg
Number analyzed (Participants) | 34 | 26
Months | 1.885 [1.541 to 3.738] | 2.148 [1.016 to 7.344]

7. Post Hoc Outcome: Median Overall Survival (OS) in Treatment With Intrathecal Trastuzumab for Patients With Leptomeningeal Metastases in HER2+ Breast Cancer.
Description: Overall Survival (OS) will be measured from start of treatment until death from any cause. To estimate OS, Kaplan-Meier curves will be calculated and median OS will be determined from the progression-free survival curve.
Time Frame: From start of treatment until death from any cause for up to 60 months.
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment With Trastuzumab | Cohort 5 + Phase II - Intrathecal Trastuzumab- 80 mg
Number analyzed (Participants) | 34 | 26
percentage of patients | 8.738 [5.607 to 17.311] | 8.328 [5.148 to 19.541]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 6 year period for the study. Patients were followed from first day of treatment until 30 days post first treatment for a maximum of 22 cycles (longest time any patient received treatment) where 1 cycle = 28 days.
Arm/Group | Cohort 1 - Trastuzumab 10mg IT 2/Week | Cohort 2 - Trastuzumab 20mg IT 2/Week | Cohort 3- Trastuzumab 40mg IT 2/Week | Cohort 4 - Trastuzumab 60mg IT 2/Week | Cohort 5 - 80mg IT 2/Week | Phase II - Transtuzumab 80mg IT 2/Week
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 1/1 | 1/1 | 5/7 | 17/19
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/1 | 1/1 | 3/7 | 13/19
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1 | 1/1 | 7/7 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Trastuzumab 10mg IT 2/Week (N=3) | Cohort 2 - Trastuzumab 20mg IT 2/Week (N=3) | Cohort 3- Trastuzumab 40mg IT 2/Week (N=1) | Cohort 4 - Trastuzumab 60mg IT 2/Week (N=1) | Cohort 5 - 80mg IT 2/Week (N=7) | Phase II - Transtuzumab 80mg IT 2/Week (N=19)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient also experienced venous thromboembolism during inpatient hospitalization.
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chemical meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Worsening Mental Status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal muscle wall hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient experienced abdominal pain during this event.
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death due to aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Patients experienced generalized weakness and abdominal pain during the inpatient hospitalization.
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasivagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient experienced nausea during this inpatient hospitalization.
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient also experienced confusion during this inpatient hospitalization.
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (DVT) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient also experienced pulmonary embolism during this inpatient hospitalization.
Death due to progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in back and extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient also experienced Nausea and headache during this inpatient hospitalization
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clinical deterioration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Worsening neurological symptoms (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Patient also experienced gait disturbance during this hospitalization.
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Patient also experienced somnolence during this hospitalization.
Arachnoiditis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Trastuzumab 10mg IT 2/Week (N=3) | Cohort 2 - Trastuzumab 20mg IT 2/Week (N=3) | Cohort 3- Trastuzumab 40mg IT 2/Week (N=1) | Cohort 4 - Trastuzumab 60mg IT 2/Week (N=1) | Cohort 5 - 80mg IT 2/Week (N=7) | Phase II - Transtuzumab 80mg IT 2/Week (N=19)
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 4 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 3 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 3
Decreased appetite (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Edema in limbs (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Edema in head (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 3 | 4
Fever (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 1 | 2 | 5
Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 1 | 3 | 3
Blood Antidiuretic Hormone Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 2 | 0 | 0 | 0 | 1 | 8
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 5
White Blood Cell Decreased (Investigations) | 1 | 1 | 0 | 0 | 1 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 4 | 4
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 3 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 2 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 5 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abducens Nerve Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headaches (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 3
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Meningismus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Involuntary Movements (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oculomotor Nerve Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gait difficulty (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2
Urinary Frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hand and Foot Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hematuria (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 6 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hot Flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic Event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes